CLINICAL TRIAL: NCT00364611
Title: A Pilot, Phase II, Multicenter, Open-Label, Prospective Evaluation of Docetaxel and Bevacizumab ± Trastuzumab in the First-Line Treatment of Patients With Metastatic Breast Cancer
Brief Title: Pilot Study of Docetaxel & Bevacizumab +/- Trastuzumab in First-Line Treatment of Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_00712
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Trastuzumab

ARMS (2):
- Docetaxel and Bevacizumab (Experimental): Stratum 1: HER2 Negative participants with metastatic breast cancer treated with DB (docetaxel and bevacizumab) intravenously (IV) every 3 weeks (q3w) until treatment discontinuation criteria (unacceptable toxicity, disease progression or death) are met
  Interventions: Drug: Bevacizumab; Drug: Docetaxel
- Docetaxel, Bevacizumab and Trastuzumab (Experimental): Stratum 2: HER2 Positive participants with metastatic breast cancer treated with DBT (docetaxel, bevacizumab, and trastuzumab) IV q3w until treatment discontinuation criteria (unacceptable toxicity, disease progression or death) are met
  Interventions: Drug: Bevacizumab; Drug: Docetaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (Avastin) 15 mg/kg will be administered prior to chemotherapy on
  * On Day 1 of the 1st cycle over 120 minutes
  * On Day 1 of the 2nd cycle over 90 minutes, if no reaction on the first dose
  * On Day 1 of 3rd cycle over 60 minutes, if no reaction on previous doses
  * On Day 1 of subsequent cycles over 30 minutes, if no reaction on previous doses
  Other Names: Avastin
Drug: Docetaxel — Docetaxel 75 mg/m^2 IV infused over 60 minutes after completion of Bevacizumab infusion q3w
Drug: Trastuzumab — * A loading dose of 8 mg/kg Trastuzumab (Herceptin) IV will be infused over 90 minutes on Day 2 of Cycle 1.
  * For all subsequent cycles 6 mg/kg trastuzumab will be administered on Day 1 one hour following completion of docetaxel infusion
  Other Names: Herceptin
  Arms: Docetaxel, Bevacizumab and Trastuzumab

SUMMARY:
Pilot, phase II, parallel-group, open-label, noncomparative, prospective, multicenter study designed to evaluate the progression-free survival of docetaxel and bevacizumab ± trastuzumab for the first-line treatment of participants with metastatic breast cancer. Participants were stratified according to human epidermal growth factor receptor-2 (HER2) status at the time of enrollment. HER2 negative participants were assigned to receive docetaxel and bevacizumab (DB). HER2 positive participants were assigned to receive docetaxel, bevacizumab, and trastuzumab (DBT).

All participants (except one) were off study treatment on 30 June 2011. All efficacy analysis and safety analysis was performed using the cut-off date of June 2011. One participant continued treatment till 11 March 2012. For this participant, adverse events were collected upto 19 April 2012 and included in the safety analysis.

DETAILED DESCRIPTION:
The study included:

* Study registration on Day 1: Treatment Cycle 1 was initiated within 14 days of signing informed consent
* Treatment was administered in 3 week treatment cycles until the participant developed unacceptable toxicity, had disease progression, withdrew consent, or died
* If participants experienced a complete response (CR), partial response (PR), or stable disease (SD) at Cycle 8 or beyond or had unacceptable toxicity due to docetaxel, they could continue on bevacizumab and/or trastuzumab until they developed unacceptable toxicity, had disease progression, or withdrew consent
* Participants had follow-up assessments within 30 days after discontinuation of treatment with the last of the study drugs for any reason other than death

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow participants and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

INCLUSION CRITERIA:

1. Histologically or cytologically proven adenocarcinoma of the breast at first diagnosis
2. Stage IV disease with at least one measurable lesion according to the RECIST criteria
3. HER2/neu positive as determined by 3+ immunohistochemistry (IHC) staining or fluorescence in situ hybridization (FISH) positivity or negative tumors
4. Life expectancy of >/= 24 weeks
5. No prior chemotherapy for metastatic breast cancer. (Prior endocrine therapy is permitted).
6. Prior neoadjuvant or adjuvant chemotherapy is permitted, or at least 12 months must have elapsed since the neoadjuvant or adjuvant therapy. Subjects may have received prior adjuvant anthracyclines (maximum cumulative dose, 360 mg/m^2 doxorubicin or 750 mg/m^2 epirubicin)
7. At least 4 weeks since prior surgery, radiotherapy, endocrine therapy, or experimental drug therapy with complete recovery from the effects of these interventions
8. It is recommended that all baseline staging should be completed within 35 days prior to study entry. All subjects will have the following workup as applicable; CT scan of brain, CT scan or MRI of chest and abdomen, and bone scan or PET scan. In cases of positive bone or PET scans, bone X-ray evaluation and/or MRI is required to confirm or exclude metastatic bone disease. Subjects with metastatic disease limited to bone are ineligible unless at least one lytic lesion is measurable and can be followed by RECIST criteria. Other tests may be performed as clinically indicated
9. Normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF) of >/= 50% or shortening fraction (multiple-gated acquisition [MUGA] scan or echocardiography respectively). The result must be greater than the lower limit of normal (LLN) for the institution.
10. Subjects receiving bisphosphonate therapy; however, if bisphosphonates were started within <2 months prior to treatment the bone lesions will not be evaluated for response, and the subjects must have another site of metastatic disease that is either measurable or evaluable for response

EXCLUSION CRITERIA:

1. Prior chemotherapy for metastatic breast cancer
2. Prior treatment with bevacizumab or other anti-VEGF therapy
3. Concurrent treatment with any other non-protocol anticancer therapy with the exception of radiation therapy as long as all target lesions being followed are not in the radiation field and if HER2/neu positive, HER2/neu-directed therapy
4. Current or prior history of brain or leptomeningeal metastases
5. Presence of neuropathy >/= 2
6. Presence of any non-healing wound, fracture, or ulcer, or the presence of clinically significant (>/= Grade 2) peripheral vascular disease
7. History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma in-situ of the cervix
8. Clinically significant cardiovascular disease
9. Active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to beginning therapy
10. History of bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-08; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Childs, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 participants signed the informed consent for this study. Of these, 73 were determined to be eligible for inclusion. One participant did not receive any study treatment.
Period: Overall Study
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Started | 52 | 21
TREATED (SAFTEY POPULATION) | 52 (Received at least one dose of study medication) | 20 (Received at least one dose of study medication)
Completed | 1 (Ongoing treatment (June 2011-initial analysis). Continued treatment till March 2012 (study closed).) | 0
Not Completed | 51 | 21
Not completed — Did not receive study medication | 0 | 1
Not completed — Adverse Event | 7 | 4
Not completed — Participant's Request | 3 | 4
Not completed — Disease Progression | 38 | 8
Not completed — Investigator decision | 2 | 2
Not completed — Found Ineligible | 1 | 0
Not completed — Presumed CR on Study | 0 | 1
Not completed — Receiving Liver Ablation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab | Total
Number analyzed (Participants) | 52 | 21 | 73
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.78) | 52.8 (12.65) | 55.2 (11.37)
Age, Customized [Number; unit: participants]
  <=65 years | 41 | 17 | 58
  Between 65 and 75 years | 8 | 3 | 11
  >=75 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 21 | 73
  Male | 0 | 0 | 0
Eastern Cooperative Oncology [Number; unit: participants] — The ECOG performance status score is used to assess how a patient's disease is progressing and to assess how the disease affects the patient's daily living abilities. The ECOG score ranges from 0-5, with 0 indicating the best outcome and a score of 5 indicating the worst outcome. An ECOG score "0" reflects a fully active patient, able to carry on all pre-disease performance without restriction. An ECOG score "1" reflects a participant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  participants
    ECOG Performance Score is 0 | 28 | 16 | 44
    ECOG Performance Score is 1 | 24 | 5 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate: Percentage of Participants With PFS
Description: PFS was the time from registration to first documentation of
  * progressive disease (PD) based on Response Evaluation Criteria in Solid Tumors (RECIST) - criteria pre-defining changes in lesion size or appearance
  * symptomatic deterioration
  * death due to any cause (in absence of PD).
  The Percentage of participants with PFS is reported.
  For the analysis, participants were censored
  * on the last available tumor assessment date on study treatment if they
    * had no PFS event
    * were on anticancer therapy not related to study treatment
  * on the registration date if they
    * did not receive study drug
    * had no post baseline tumor assessment
Time Frame: Up to 6 months and 12 months after treatment initiation
Population: Intent to treat population: all registered participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Number analyzed (Participants) | 52 | 21
percentage of participants
  PFS rate at 6 months | 59.6 [45.1 to 73.0] | 90.5 [69.6 to 98.8]
  PFS rate at 12 months | 30.8 [18.7 to 45.1] | 81.0 [58.1 to 94.6]

2. Primary Outcome: Time to Progression-free Survival (PFS)
Description: Time to PFS was the interval from the date of registration to the earliest of the following documented dates:
  * PD as defined by RECIST (criteria pre-defining changes in lesion size or appearance)
  * symptomatic deterioration
  * death.
  Time to PFS was estimated from Kaplan-Meier Plots.
Time Frame: From treatment initiation to PFS event (up to June 2011)
Population: Intent-to-treat population: all registered participants
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: PFS events analyzed
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Number analyzed (Participants) | 52 | 21
Number analyzed (PFS events analyzed) | 45 | 10
days | 255 [158 to 315] | 403 [363 to 1078]

3. Secondary Outcome: Confirmed Overall Response (OR) Based on RECIST Criteria
Description: Confirmed OR was confirmed Complete Response (CR) + confirmed Partial Response (PR). According to RECIST
  * CR was the disappearance of all tumor lesions
  * PR was a pre-defined decrease in the size of tumor lesions.
  To determine a response, radiologic tumors assessments were performed using computed tomography (CT) and/or magnetic resonance imaging (MRI) of the chest, and the abdomen, bone scan or positron emission tomography (PET) scan, and other imaging techniques as clinically indicated. To confirm a response, 2 assessments separated by 28 days or more were required.
Time Frame: From treatment initiation to June 2011
Population: Intent-to-treat population: all registered participants.
Measure: Number; unit: participants
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Number analyzed (Participants) | 52 | 21
participants
  Confirmed overall response | 30 | 17
  Confirmed complete response | 3 | 4
  Confirmed partial response | 27 | 13

4. Secondary Outcome: Number of Participants With Confirmed Clinical Benefit Based on RECIST Criteria
Description: Clinical Benefit (CB) was achieved in participants with a response (CR + PR) or a stable disease (SD).
  According to RECIST
  * CR was the disappearance of all tumor lesions
  * PR was a pre-defined decrease in the size of tumor lesions
  * SD was neither sufficient decrease in tumor size to qualify for PR or sufficient increase to qualify for PD.
  Confirmation of a response needed 2 responses scored, separated by 28 days or more (for CR and PR), and by 26 weeks or more (for SD).
Time Frame: From treatment initiation to June 2011
Population: Intent-to-treat: all registered participants.
Measure: Number; unit: participants
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Number analyzed (Participants) | 52 | 21
participants
  with confirmed Clinical Benefit (CR+PR+SD) | 35 | 17
  with confirmed CR | 3 | 4
  with confirmed PR | 27 | 13
  with confirmed SD | 14 | 1

5. Secondary Outcome: Duration of Response (DR)
Description: DR was the interval from date of initial documented confirmed response (CR or PR) to the first documented confirmed date of disease progression (PD) or death from any cause in the absence of previous documentation of objective tumor progression.
  Participants who were alive and without any record of PD at the time of discontinuation were censored at the last available tumor assessment date; participants with non-study anti-cancer therapy during the study were censored at the last available tumor assessment date prior to the anti-cancer therapy.
  DR was estimated from Kaplan-Meier Plots.
Time Frame: From treatment initiation to June 2011
Population: Participants with a documented response of CR or PR.
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Events (PD or death after 1st Response)
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Number analyzed (Participants) | 30 | 17
Number analyzed (Events (PD or death after 1st Response)) | 25 | 8
days | 232 [126 to 305] | 366 [293 to 859]

6. Secondary Outcome: Overall Survival (OS) Time
Description: OS was the interval between the date of study entry and the date of death from any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive.
  OS time was estimated from Kaplan-Meier Plots.
Time Frame: From treatment initiation to June 2011
Population: Intent-to-treat population: all registered participants.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Deaths
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Number analyzed (Participants) | 52 | 21
Number analyzed (Deaths) | 33 | 6
days | 750 [362 to 1159] | 986 [619 to 1705]

7. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An adverse event (AE) was any unfavorable and unintended sign, symptom, syndrome, or illness that developed or worsened during the clinical study. AEs occurring on or after first dose of study medication inclusive to 30 days post-last dose were the treatment emergent adverse events (TEAEs).
  An serious adverse event was an AE that at any dose (including overdose) resulted in death, was life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly, and/or was medically important.
Time Frame: From treatment initiation to 30 days after the last dose of study treatment
Population: Safety population: all participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Number analyzed (Participants) | 52 | 20
participants
  with treatment emergent adverse events (TEAEs) | 52 | 20
  with serious adverse events | 14 | 4
  with TEAEs resulting in death | 3 | 0

ADVERSE EVENTS:
Time Frame: From treatment initiation up to 30 days following the last dose of study medication (upto April 2012)
Description: All participants (except one) were off study treatment on 30 June 2011. An initial safety analysis was performed using the cut-off date of June 2011. One participant continued till 19 April 2012. For this participant, adverse events were collected upto April 2012 and included in the final safety analysis.
Arm/Group | Docetaxel and Bevacizumab | Docetaxel, Bevacizumab and Trastuzumab
Serious Adverse Events (participants affected / at risk) | 14/52 | 4/20
Other Adverse Events (participants affected / at risk) | 52/52 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and Bevacizumab (N=52) | Docetaxel, Bevacizumab and Trastuzumab (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and Bevacizumab (N=52) | Docetaxel, Bevacizumab and Trastuzumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Tachycardia (Cardiac disorders) | 3 | 1
Lacrimation increased (Eye disorders) | 15 | 10
Dry eye (Eye disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 28 | 10
Diarrhoea (Gastrointestinal disorders) | 23 | 8
Constipation (Gastrointestinal disorders) | 17 | 4
Vomiting (Gastrointestinal disorders) | 12 | 7
Stomatitis (Gastrointestinal disorders) | 9 | 6
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2
Fatigue (General disorders) | 36 | 13
Mucosal inflammation (General disorders) | 14 | 3
Oedema peripheral (General disorders) | 12 | 3
Pain (General disorders) | 5 | 2
Pyrexia (General disorders) | 5 | 2
Chills (General disorders) | 4 | 1
Chest pain (General disorders) | 3 | 0
Asthenia (General disorders) | 1 | 3
Urinary tract infection (Infections and infestations) | 9 | 6
Sinusitis (Infections and infestations) | 8 | 5
Furuncle (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Nail infection (Infections and infestations) | 3 | 4
Nasopharyngitis (Infections and infestations) | 1 | 2
Eye infection (Infections and infestations) | 0 | 2
Weight decreased (Investigations) | 8 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood creatinine increased (Investigations) | 3 | 0
Ejection fraction decreased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 10 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 20 | 8
Headache (Nervous system disorders) | 16 | 9
Neuropathy peripheral (Nervous system disorders) | 11 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 4
Dizziness (Nervous system disorders) | 6 | 1
Memory impairment (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 10 | 5
Anxiety (Psychiatric disorders) | 7 | 4
Depression (Psychiatric disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 7 | 3
Dysuria (Renal and urinary disorders) | 4 | 0
Breast pain (Reproductive system and breast disorders) | 4 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 15
Nail disorder (Skin and subcutaneous tissue disorders) | 18 | 7
Erythema (Skin and subcutaneous tissue disorders) | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 2
Sinus operation (Surgical and medical procedures) | 1 | 2
Hypertension (Vascular disorders) | 7 | 8
Hot flush (Vascular disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 60 days in advance of any submission for publication. The Sponsor may request for the publication to be delayed for a limited time, not to exceed 90 days to preserve its proprietary rights.